CLINICAL TRIAL: NCT05930496
Title: A Randomized Controlled Trial Testing the Effects of an Exercise Intervention on the Gut Microbiota in Colorectal Cancer Survivors: A Pilot and Feasibility Study
Brief Title: Evaluating the Effects of an Exercise Intervention on the Gut Microbiota in Stage II-III Colorectal Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1123467; NCI-2023-03747 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH); 20059 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Stage II Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Specimen Handling; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (exercise intervention) (Experimental): Patients receive the supervised exercise intervention over 8 weeks on study. Patients also undergo collection of blood samples at baseline and week 8.
  Interventions: Procedure: Biospecimen Collection; Other: Exercise Intervention; Other: Interview; Other: Questionnaire Administration
- Arm B (waitlist control) (Active Comparator): Patients receive health-related information for 8 weeks on study. Patients are then offered a session of supervised exercise followed by 7 weeks of tele-coaching sessions. Patients also undergo collection of blood samples at baseline and week 8.
  Interventions: Procedure: Biospecimen Collection; Other: Exercise Intervention; Behavioral: Health Education; Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Exercise Intervention — Receive exercise intervention
  Arms: Arm A (exercise intervention)
Other: Exercise Intervention — Receive tele-coaching intervention
  Arms: Arm B (waitlist control)
Behavioral: Health Education — Receive health-related information
  Arms: Arm B (waitlist control)
Other: Interview — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial evaluates the effects a moderate-to-vigorous exercise intervention has on the bacterial make-up of the gastrointestinal tract (gut microbiota) in survivors of stage II-III colorectal cancer (CRC). Data shows that the gut microbiota composition and function may be drivers of CRC. High levels of exercise are associated with improved CRC prognosis and survival. While data suggests that exercise has the potential to influence gut microbiota composition and function, it is not known whether these effects contribute to improved CRC prognosis. This clinical trial evaluates the effects an exercise intervention has on gut microbiota and how these effects relate to CRC progression and patient-reported outcomes.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive the supervised exercise intervention over 8 weeks on study. Patients also undergo collection of blood samples on study.

ARM B: Patients receive health-related information for 8 weeks on study. Patients are then offered a session of supervised exercise followed by 7 weeks of tele-coaching sessions. Patients also undergo collection of blood samples on study.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Previous diagnosis of stage II-III CRC cancer
* No known current, recurrent, or metastatic disease
* No comorbid or physical limitations that would limit participation at the discretion of the treating provider
* At least 60 days to 3 years from last cancer-directed treatment (including surgery, chemotherapy, and radiation. Elective surgery, including ileostomy reversal, is not counted in this timing but patients must be able to eat a normal diet, without post-operative dietary limitations)
* Body mass index (BMI) 18.5-30 kg/m^2
* Able to understand and willing to sign written informed consent in English
* Access to phone for study contacts
* Be willing and able to attend the 24 sessions at the Fred Hutch Exercise Research Center Shared Resource
* Access to internet
* Willingness to participate in all study activities
* Completion of all run-in activities
* Participants must not be active smokers within the past 30 days. Active smoking is defined as any smoking (of cigarettes or tobacco products), even a puff

  * Participants who smoke are much less likely to engage in healthy lifestyle behaviors, and it is probably more important for participants to stop smoking than it is to change their exercise patterns. If identified as a smoker, the individual will be referred to the local resources, Washington State Quitline (1-800-QUIT-NOW), ICanQuit.org, Quit2Heal.org, the national resource, Centers for Disease Control and Prevention (CDC) "Quit Now" phone line which supports smoking cessation, or the National Institutes of Health (NIH) quit support website "SmokeFree.gov"
* At time of consent, participants must engage =< 60 minutes per week of moderate to vigorous physical activity, as assessed by brief questionnaires at screening and then objectively assessed using accelerometers at baseline
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Scale of Performance Status score of 0 or 1 for performance status
* Physician approval for participation in an 8-week exercise program
* Women must not be pregnant, breastfeeding, or planning to become pregnant

Exclusion Criteria:

* Use of oral or intravenous antibiotics, antifungals, or antiparasitics during the past 6 months
* Presence of an ileostomy or colostomy because of known changes to the gut microbiome with ileostomies and colostomies
* Current status of underweight (BMI < 18.5 kg/m^2) or obese (BMI >= 30.0 kg/m^2)
* Presence of inflammatory bowel diseases such as Crohn's disease or ulcerative colitis as these are known to baseline have differences in gut microbiome composition
* Active smokers within the past 30 days
* Women who are pregnant, breastfeeding, or planning to become pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Up to 8 weeks
  Recruitment (accrual rate) will be assessed to determine feasibility. Will be summarized using descriptive statistics.
Adherence | Up to 8 weeks
  Adherence will be measured by session attendance in the intervention arm to determine feasibility. Will be summarized using descriptive statistics.
Retention | Up to 8 weeks
  Retention will be measured by completion of all study assessments, including physical activity via accelerometry, 24 hour dietary recalls, and completion of the follow-up data collection at 8 weeks to determine feasibility. Will be summarized using descriptive statistics. Statistical differences in retention rates for each study assessment between study arms will be assessed by logistic regression models and acceptability by linear regression models, with models adjusted for stratification factors.
Acceptability | Up to 8 weeks
  Acceptability will be measured on a Likert scale in each of a series of questions regarding various aspects of the trial during the exit interview to determine feasibility. Will be summarized using descriptive statistics.

SECONDARY OUTCOMES:
Effects of an 8 week supervised exercise intervention on fecal concentrations of butyrate | At 8 weeks
  Will be summarized using descriptive statistics, and statistical differences between study arms will be assessed via linear regression models with adjustment for baseline outcome values and stratification factors.
Effects of an 8 week supervised exercise intervention on fecal concentrations of other short chain fatty acids | At 8 weeks
  Will be summarized using descriptive statistics, and statistical differences between study arms will be assessed via linear regression models with adjustment for baseline outcome values and stratification factors.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Greenlee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No